CLINICAL TRIAL: NCT00940589
Title: A Double-blind, Parallel Group, Randomized, Placebo Controlled Study of the Efficacy of Circadin® 2mg in Patients With Mild to Moderate Alzheimer Disease (AD) Treated With Acetylcholinesterase (AChE) Inhibitor
Brief Title: Efficacy of Circadin® 2 mg in Patients With Mild to Moderate Alzheimer Disease Treated With AChE Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEU AZ1
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Alzheimer's Disease; Sleep Disorder
Keywords: Alzheimer's Disease; Acetylcholinesterase inhibitor; cognitive function; Circadin; Sleep disturbances
MeSH Terms: conditions — Alzheimer Disease; Sleep Wake Disorders; Parasomnias | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circadin (Experimental): Drug
  Interventions: Drug: Circadin
- Placebo (Placebo Comparator): drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Circadin — Prolonged Release melatonin (Circadin) 2mg tablets
  Arms: Circadin
Drug: Placebo — Matched placebo tablets, with identical features to the Circadin tablets
  Arms: Placebo

SUMMARY:
The aim of this exploratory randomized, placebo controlled study is to evaluate the efficacy of Circadin® 2mg in patients with mild to moderate Alzheimer Disease (AD) treated with the acetylcholinesterase (AChE) inhibitor. The effects of add-on Circadin® 2mg vs. placebo on the decline in cognitive skills and global functioning, as well as on daytime somnolence and will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent as dictated by local legal circumstances.
2. Age range: adult patients between 50-85 years of age.
3. Gender: men and women. Women of child bearing potential or within two years of the menopause must have a negative urine pregnancy test at the Screening Visit.
4. A documented history of confirmed Alzheimer's disease
5. Dementia severity: MMSE score > 15,
6. Stable AChE inhibitor dose for 2 months prior to Screening visit.
7. Stable medications for non-excluded concurrent medical conditions for four weeks prior to the screening visit.
8. Stable doses of B12 and/or Folic acid supplements for at least 3 months prior to enrollment and throughout the study.
9. Cranial image: no evidence of focal disease to account for dementia (established by CT, PET or MRI). If there is no such available scan (CT, PET or MRI), one must be performed prior to enrollment.
10. Health: Physically acceptable for the study with no pathology likely to occur during or immediately after the study, as confirmed by medical history and exam and ECG.
11. Clinical laboratory values must be within normal limits, or judged not clinically significant by the investigator.
12. Residence: Stable home situation with no planned move during the 28-week investigational period.
13. A family member or a regular caregiver that will be available for visits and will ensure compliance. The caregiver must speak fluent Hebrew, Russian or English.
14. Ability to ingest oral medication and participate in all scheduled evaluations.
15. Ability to spend 2 daily hours outdoors exposed to sunlight.

Exclusion Criteria:

1. Severe agitation.
2. Unstable medical condition, mental retardation.
3. moderate to severe depression as defined by DSM-IV
4. Use of benzodiazepines or other hypnotics during the study and the preceding four weeks.
5. Use of Circadin® during the two weeks prior to study enrollment.
6. Pharmacological immunosuppression.
7. Participation in a clinical trial with any investigational agent within two months prior to study enrollment.
8. Alcoholism.
9. Known or suspected hypersensitivity to exogenous melatonin or melatonin receptor agonists.
10. Patients with rare hereditary problems of galactose intolerance, the LAPP lactose deficiency or glucose mal absorption.
11. Renal Failure with creatinine >150 micromol/l.
12. Hepatic Failure with ASAT; ALAT; GGT levels above three times the upper normal limit.
13. Clinically significant abnormal laboratory findings which have not been approved by the Safety Officer (sponsor)
14. Other serious diseases that could interfere with patient assessment.
15. Caregivers who are unwilling or unable to give informed consent or otherwise fulfill requirements of the study.
16. Untreated B12 and/or Folic acid deficiency.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Meridien Research, Brooksville, Florida
  - Meridien Research, St. Petersburg, Florida
  - Exodon LLC, Mount Arlington, New Jersey
  - Scranton Medical Institute, Scranton, Pennsylvania
- Merchav clinics, Tel Aviv, Israel
- CPS Research, Glasgow, United Kingdom

REFERENCES:
- [Result] Wade AG, Farmer M, Harari G, Fund N, Laudon M, Nir T, Frydman-Marom A, Zisapel N. Add-on prolonged-release melatonin for cognitive function and sleep in mild to moderate Alzheimer's disease: a 6-month, randomized, placebo-controlled, multicenter trial. Clin Interv Aging. 2014 Jun 18;9:947-61. doi: 10.2147/CIA.S65625. eCollection 2014. PMID 24971004
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Circadin | Placebo
Started | 39 | 34
Completed | 31 | 29
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Circadin | Placebo | Total
Number analyzed (Participants) | 39 | 34 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (8.6) | 77.3 (6.6) | 75.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 23 | 14 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Weeks in ADAS-cog
Description: ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale) is a cognitive testing instrument used in clinical trials. It consists of 11 tasks measuring the disturbances of memory, language, praxis, attention, and other cognitive abilities that are often referred to as the core symptoms of AD. The test comprises 11 items summed to a total score ranging from 0 to 70, with lower scores indicating less severe impairment. A negative change indicates an improvement from baseline. ADAS-cog was measured at base line and at end of treatment after 24 weeks.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Circadin | Placebo
Number analyzed (Participants) | 29 | 26
Scores on a scale | 0.45 (5) | 0.19 (6.28)

2. Secondary Outcome: Change From Baseline to 24 Weeks in iADL
Description: Instrumental Activities of Daily Living (iADL). The scale rates activities that represent key life tasks that people need to manage. These tasks are valuable for evaluating persons with early-stage disease, both to assess the level of disease and to determine the person's ability to care for himself or herself. Scores of 0 or 1 are given to every task (Bathing, Dressing, Tolieting, transferring, Continence and Feeding) to a total score of 6. , while 0 represents a patient who is very dependent and 6 represents patient who is independent. iADL was measured at base line and at end of treatment after 24 weeks.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Circadin | Placebo
Number analyzed (Participants) | 31 | 29
Scores on a scale | 0.77 (1.41) | 1.62 (1.57)
Statistical Analysis 1: Comparison: Circadin vs Placebo; Test type: Superiority or Other; p < 0.045, ANCOVA

3. Secondary Outcome: Change From Baseline to 24 Weeks in MMSE
Description: The Mini Mental State Examination (MMSE) is a brief assessment instrument used to assess cognitive function in elderly patients. The MMSE can be used to screen for cognitive impairment and as a measurement of cognition over time and with pharmacologic treatment. The instrument is divided into 2 sections. The first section measures orientation, memory, and attention: the maximum score is 21. The second section tests the ability of the patient to name objects, follow verbal and written commands, write a sentence, and copy figures: the maximum score is 9. The scoring range for the MMSE is 0-30. Higher score represents better performance. MMSE was measured at base line and at end of treatment after 24 weeks.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Circadin | Placebo
Number analyzed (Participants) | 32 | 29
Scores on a scale | -0.3 (2.8) | -1.9 (3.5)
Statistical Analysis 1: Comparison: Circadin vs Placebo; Test type: Superiority or Other; p < 0.044, ANCOVA

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Circadin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/39 | 5/34
Other Adverse Events (participants affected / at risk) | 32/39 | 23/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circadin (N=39) | Placebo (N=34)
esophageal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not related to the study drug.
Severe miocardial infraction (Cardiac disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Endocrine disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circadin (N=39) | Placebo (N=34)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Blood creatinine increased (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Blood glucose increased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Abnormal dreams (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2)
Cognitive disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days